CLINICAL TRIAL: NCT01074125
Title: A 4-Week Dose-Ranging and Efficacy Trial of KRX-0502 (Ferric Citrate) in Patients With End-Stage Renal Disease (ESRD) Following a Two-Week Washout Period
Brief Title: A 4-Week Dose-Ranging and Efficacy Trial of KRX-0502 (Ferric Citrate) in Patients With End-Stage Renal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Collaborators: Collaborative Study Group (CSG) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRX-0502-305
Record Dates: First submitted 2010-02-17; First posted 2010-02-24 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Hyperphosphatemia; End-Stage Renal Disease
Keywords: Hyperphosphatemia; ESRD; Dialysis; End Stage Renal Disease; Phosphorus; Renal; Kidney
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic | interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 g/day (Experimental): 1 g/day KRX-0502 (ferric citrate)
  Interventions: Drug: ferric citrate
- 6 g/day (Experimental): 6 g/day KRX-0502 (ferric citrate)
  Interventions: Drug: ferric citrate
- 8 g/day (Experimental): 8 g/day KRX-0502 (ferric citrate)
  Interventions: Drug: ferric citrate

INTERVENTIONS:
Drug: ferric citrate — 1, 6, or 8 g/day taken within 1 hour of meals or snacks daily for 28 days
  Other Names: KRX-0502

SUMMARY:
This is a research study for people with high blood phosphorus levels who are on dialysis. This medical condition can cause weakening of the bones and damage other organs. This can lead to many health problems, and sometimes death. Phosphorus is in much of the food we eat, and is helpful to us in small amounts. Patients with kidney failure have trouble getting rid of the phosphorus eaten in food. Dialysis can help remove some of the phosphorus, but often patients must take a phosphate binder like PhosLo®, Renagel®, or Renvela® to bring the blood phosphorus levels back to normal. The purpose of this study is to see if KRX-0502 (ferric citrate) is safe and effective as a phosphate binder.

DETAILED DESCRIPTION:
There will be a screening visit about 4 weeks receiving study drug. Upon qualifying for the study after the screening visit, patients will then be asked to stop taking their current phosphate binder for about 2 weeks. Then, if patients continue to qualify for the study, they will be entered in the study that lasts about 28 days. Study visits will happen every week during the patient's usual dialysis appointments. There will be a total of up to 9 visits for this study, and total participation time could last up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating females
* Age > 18 years
* On thrice weekly hemodialysis or peritoneal dialysis for at least the previous three months prior to Screening Visit (Visit 0)
* Serum phosphorus levels ≥ 3.5 mg/dL and < 8.0 mg/dL at Screening Visit (Visit 0)
* Serum phosphorus levels > 6.0 mg/dL during the washout period (Visits 2 or 3)
* Taking 3 to 15 tablets/capsules per day of 667mg calcium acetate or 800 mg sevelamer (hydrochloride or carbonate), or any combination of these agents as reported by the patient at Screening Visit (Visit 0)
* Serum ferritin <1000micrograms/L and Transferrin Saturation (TSAT) <50% at the Screening Visit (Visit 0)
* Willingness to be discontinued from current phosphate binder(s) and initiated on KRX-0502 (ferric citrate)
* Willing and able to give informed consent
* Willing and able to stay on a constant dose of Vitamin D (or its analogs) and Sensipar (cinacalcet) for the treatment period, if applicable.

Exclusion Criteria:

* Parathyroidectomy within six months prior to Screening Visit (Visit 0)
* Actively symptomatic gastrointestinal bleeding or inflammatory bowel disease
* Serum phosphorus levels >10.0 mg/dL documented in all of the three monthly laboratories (done routinely in the dialysis unit) in the three months prior to the Screening Visit (Visit 0)
* History of multiple drug allergies or intolerances
* History of malignancy in the last five years (treated cervical or non-melanomatous skin cancer may be permitted if approved by CCC)
* Previous intolerance to oral ferric citrate
* Absolute requirement for oral iron therapy
* Absolute requirement for Vitamin C (multivitamins [Nephrocaps, Renaphro, etc.] allowed)
* Absolute requirement for calcium-, magnesium-, or aluminum-containing drugs with meals
* Psychiatric disorder that interferes with the patient's ability to comply with the study protocol
* Inability to tolerate oral drug intake
* Planned surgery or hospitalization during the trial (scheduled outpatient access surgery allowed)
* Any other medical condition that renders the patient unable to or unlikely to complete the trial or that would interfere with optimal participation in the trial or produce significant risk to the patient
* Receipt of any investigational drug within 30 days of Screening Visit (Visit 0)
* Inability to cooperate with study personnel or history of noncompliance
* Unsuitable for this trial per Principal Investigator's clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia B Lewis, MD, Study Chair — Collaborative Study Group (CSG)
Locations (16):
- United States (15):
  - Western Nephrology, Westminster, Colorado
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Kidney Care Associates, LLC, Augusta, Georgia
  - Circle Medical Management, Chicago, Illinois
  - Western New England Renal & Transplant Associates, Springfield, Massachusetts
  - Brookdale Physician's Dialysis Associates, Brooklyn, New York
  - DCI, Cincinnati, Ohio
  - Cleveland Clinical Foundation Fresenius East (Fairhill), Cleveland, Ohio
  - The Ohio State University Cramblett Medical Clinic, Columbus, Ohio
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Nephrology Associates, PC, Nashville, Tennessee
  - Meharry Medical College Clinical Research Center, Nashville, Tennessee
  - Vanderbilt University Medical Center Clinical Trials Center, Nashville, Tennessee
  - Kidney Associates, Houston, Texas
  - Centre Point Dialysis, West Allis, Wisconsin
- RCMI- Clinical Research Center Medical Sciences Campus University of Puerto Rico, Rio Piedras, PR, Puerto Rico

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Dwyer JP, Sika M, Schulman G, Chang IJ, Anger M, Smith M, Kaplan M, Zeig S, Koury MJ, Blumenthal SS, Lewis JB; Collaborative Study Group. Dose-response and efficacy of ferric citrate to treat hyperphosphatemia in hemodialysis patients: a short-term randomized trial. Am J Kidney Dis. 2013 May;61(5):759-66. doi: 10.1053/j.ajkd.2012.11.041. Epub 2013 Jan 29. PMID 23369827

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients were randomized, but withdrew before initiating study treatment
Groups:
- 1 g/Day: 1 g/day KRX-0502 (ferric citrate) taken within 1 hour of meals or snacks daily for 28 days
- 6 g/Day: 6 g/day KRX-0502 (ferric citrate) taken within 1 hour of meals or snacks daily for 28 days
- 8 g/Day: 8 g/day KRX-0502 (ferric citrate) taken within 1 hour of meals or snacks daily for 28 days
Period: Overall Study
Arm/Group | 1 g/Day | 6 g/Day | 8 g/Day
Started | 51 | 52 | 48
Completed | 39 | 47 | 36
Not Completed | 12 | 5 | 12

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 g/Day | 6 g/Day | 8 g/Day | Total
Number analyzed (Participants) | 50 | 51 | 45 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 37 | 39 | 115
  >=65 years | 11 | 14 | 6 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 19 | 58
  Male | 32 | 30 | 26 | 88
Region of Enrollment [Number; unit: participants]
  United States | 47 | 49 | 42 | 138
  Puerto Rico | 3 | 2 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphorus From Baseline to End of Treatment
Description: Mean change from baseline was calculated separately for each treatment arm (LOCF)
Time Frame: Baseline and day 28
Population: Intent to Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1 g/Day | 6 g/Day | 8 g/Day
Number analyzed (Participants) | 50 | 51 | 45
mg/dL | -0.10 (1.285) | -1.86 (1.692) | -2.13 (1.998)
Statistical Analysis 1: Comparison: 1 g/Day vs 6 g/Day vs 8 g/Day; To assess dose ranging, the primary efficacy variable will be analyzed via a model with dose effect. Positive dose ranging confirmed if the null hypothesis of slope =0 was rejected at a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = -0.3376

2. Secondary Outcome: Pairwise Comparison of the Mean Change in Serum Phosphorus From Baseline to the End of Treatment
Description: Mean change from baseline was calculated separately for each treatment arm. Only subjects that have both baseline and end of treatment serum phosphorus scores were analyzed for this outcome.
Time Frame: Baseline and day 28
Population: Intent-to-Treat, includes only subjects that had both baseline and end of study actual values
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1 g/Day | 6 g/Day | 8 g/Day
Number analyzed (Participants) | 38 | 44 | 34
mg/dL | 0.04 (1.320) | -1.94 (1.813) | -2.21 (2.097)

3. Secondary Outcome: Proportion of Patient With a Serum Phosphorus ≤5.5 mg/dL at the End of Treatment
Description: proportion was calculated separately for each treatment arm
Time Frame: Baseline and day 28
Population: Intent-to-Treat
Measure: Number; unit: % of Participants
Arm/Group | 1 g/Day | 6 g/Day | 8 g/Day
Number analyzed (Participants) | 50 | 51 | 45
% of Participants | 12.0 | 51.0 | 57.8

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (AEs) were recorded up to 30 days post therapy
Groups:
- 1g/Day: Participants received 1g tablet of KRX-0502 (ferric citrate) for 4 weeks
- 6g/Day: Participants received 6g tablet of KRX-0502 (ferric citrate) for 4 weeks
- 8g/Day: Participants received 8g tablet of KRX-0502 (ferric citrate) for 4 weeks
Arm/Group | 1g/Day | 6g/Day | 8g/Day
Serious Adverse Events (participants affected / at risk) | 6/51 | 7/52 | 9/48
Other Adverse Events (participants affected / at risk) | 34/51 | 43/52 | 41/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1g/Day (N=51) | 6g/Day (N=52) | 8g/Day (N=48)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous absess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Hypotension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 (0)
Pulmonary Odema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Renal transplant (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1g/Day (N=51) | 6g/Day (N=52) | 8g/Day (N=48)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 6 (6) | 13 (13)
Faeces discoloured (Gastrointestinal disorders) | 10 (10) | 12 (12) | 7 (7)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 9 (9)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No